CLINICAL TRIAL: NCT05492136
Title: Unravelling the Impact of Radiofrecuency in Liver Surgery: the Key to Decrease Local Recurrence? (Study LIVERaTION)
Brief Title: Unravelling the Impact of Radiofrecuency in Liver Surgery: the Key to Decrease Local Recurrence?
Acronym: LIVERaTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Patricia Sanchez Velazquez, Principal Investigator, Hospital del Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Liveration_v2
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Liver Cancer; Cancer, Treatment-Related
MeSH Terms: conditions — Liver Neoplasms; Neoplasms, Second Primary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Control (No Intervention): In this arm it will be permitted one/several conventional methods according to surgeon preference:
  * Conventional crusch-clamp or finger fracture technique
  * Ultrasonic dissector (CUSA, SONOK..) or Ultrasonic mediated devices
  * Water jet dissector
  * Argon beam coagulator
- Arm 2: study arm (Experimental): In this arm it will be permitted to use the radiofrequency devices which have demonstrated evidence in the literature in terms of reducing local recurrence alone or in combination with any conventional method described previously in Arm. (Coolingbis device by VecMedical as well as Aquamantys (Medtronic) These devices and their operating procedure have been described in detail elsewhere Briefly, it consists of a handheld instrument that might be employed not only for margin coagulation but also as hemostatic instrument. After performing the hepatectomy the bladeless part of the device should be applied onto the surgical margin following the protocol 3-4 s/cm2 of liver transection surface at maximum power output.in order to perform an additional margin coagulation
  Interventions: Procedure: Additional margin coagulation

INTERVENTIONS:
Procedure: Additional margin coagulation — After performing the hepatectomy the selected device should be applied onto the surgical margin following the protocol 3-4 s/cm2 of liver transection surface at maximum power output in order to perform an additional margin coagulation
  Arms: Arm 2: study arm

SUMMARY:
Radiofrequency devices have been increasingly employed in liver surgery in order to achieve proper hemostasis and this use has become more evident with the implementation of minimal invasive surgery. Due to its well-known efficacy for tumor ablation (i.e. hepatocarcinoma) it use has been extended in some cases to ablate the liver surface after resection in questionable resection. Till date, despite the majority of surgeons apply an additional coagulation in doubtful margins, there is not an evidence that this maneuver really decreases the local recurrence or increases the overall survival. On the contrary, some studies have suggested that non-anatomical resections in order to spare liver parenchyma could lead to major zones of liver ischemia in the remnant liver and thus favoring recurrence. However, major liver ischemia (defined as grade 2 o more) is unlikely to be provoked by 1 cm-depth additional coagulation of the margin.

The investigators previously published in a retrospective study the concept of additional margin coagulation within liver resections and narrow margins and demonstrated that the study group had significantly less local recurrence compared to the controls. Therefore, in the present study the aim is to continue this evaluation through a multicenter randomized clinical trial.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent granted prior to the initiation of the surgical procedure, given with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
2. 18 year of age or older.
3. WHO performance scale 0-2
4. Consecutive patients (both sexes equally distributed) suffering from CRLM confirmed either by abdominal CT, abdominal MRI or/and by histologic-cytological evaluation or patients suffering from HCC.
5. Any previous chemotherapy regime is permitted.
6. ASA score 1 to 3.

Exclusion criteria:

1. Previous or concurrent cancer that is distinct from one primary tumor of which the Liver metastasis comes from EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1).
2. Any cancer curatively treated > 3 years prior to enrollment is permitted.
3. ASA 4.
4. Non-resectable extrahepatic metastases.
5. Liver metastasis from other origin apart from colorectal.
6. Bening primary tumor of the liver.
7. Pregnant woman.
8. Participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Local recurrence | 5 years follow-up
  Local recurrence (LR): defined as any growing or enhancing tumour in the margin of hepatic resection specifically reviewed to this aim in a later follow-up imaging

SECONDARY OUTCOMES:
overall survival (OS) | From the surgery to death or lost of follow-up whichever came first, assessed up to 24 months
  defined as time from surgery until death or the end of the study, patients who discontinue from the study without disease will be censored at the time of their last tumour evaluation prior to death or discontinuation.
Disease free survival (DFS) | 2 years of follow-up
  Disease free survival (DFS), calculated as the time from surgery until disease progression, patients who have not progressed at the time the SVR analysis is performed will be censored at the time of their last tumour evaluation
Cancer specific survival (CSS) | From the surgery to recurrence/last follow-up whichever came first, assessed up to 24 months
  Cancer-specific survival (CSS), measured from the date of surgery to the date of death from colorectal cancer/HCC or last follow-up.
Postoperative complications | 90 days after surgery
  Graded by Clavien-Dindo clasification and CCI
Hepatic recurrence | From the surgery to hepatic recurrence or lost of follow-up whichever came first, assessed up to 24 months
  Tumoral recurrence within the liver

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Sánchez Velazquez, MD PhD FEBS, Principal Investigator — Hospital del Mar
Locations (1):
- Hospital del Mar Research Institute, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luque Villalobos E, Ielpo B, Aldrighetti L, Anselmo A, Beghdadi N, Berardi G, Briceno F, Ciria R, Dorcaratto D, Durczynski A, Ettorre GM, Delvecchio A, Ferri V, Grat M, Garces-Albir M, Grochola LF, Hogendorf P, Izzo F, Kobryn K, Kontis E, Korkolis D, Krol R, Lesurtel M, Lopez-Ben S, Christogiannis C, Koutsiouroumpa O, Mavridis D, Memeo R, Murawa D, Machairas N, Mora-Oliver I, Munoz-Forner E, Orrego C, Dantas C, Fuste C, Garcia Picazo A, Pessaux P, Pilat T, Pittau G, Radosevic A, Ratti F, Sotiropoulos G, Toutouzas K, Trotovsek B, Wystrychowski W, Zacharoulis D, Vicente E, Burdio F, Sanchez Velazquez P. LIVERATION trial: a multicentre European randomised study on radiofrequency margin coagulation and its impact on oncological outcomes after liver surgery - study protocol. BMJ Open. 2025 Nov 24;15(11):e100518. doi: 10.1136/bmjopen-2025-100518. PMID 41290310
- See also: Website — https://liveration.eu

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT05492136/SAP_000.pdf